CLINICAL TRIAL: NCT03185806
Title: A Randomized, Multicenter and Prospective Trial of Early Percutaneous Catheter Drainage of Sterile Pancreatic Fluid Collections in Severe Acute Pancreatitis
Brief Title: A Trial of Early Percutaneous Catheter Drainage of Sterile Pancreatic Fluid Collections in Severe Acute Pancreatitis
Acronym: EPCDSAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAHZhejiangU-EPCDSAP
Record Dates: First submitted 2017-05-30; First posted 2017-06-14 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2017-05

CONDITIONS: Severe Acute Pancreatitis
Keywords: severe acute pancreatitis; sterile acute peripancreatic fluid collections; percutaneous catheter drainage
MeSH Terms: conditions — Pancreatitis | interventions — Paracentesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Puncture and Drainage (Experimental): The enrolled SAP patients are administered puncture and drainage use 8-F or 10-F pigtail tube under guidance of B ultrasound or CT scan.
  Interventions: Device: Puncture and drainage
- Conservative therapy (No Intervention): The enrolled SAP patients are administered conservative therapy and without puncture and prolonged drainage.

INTERVENTIONS:
Device: Puncture and drainage — The enrolled SAP patients are punctured under guidance of B ultrasound or CT scan, and prolonged drained by 8-F or 10-F pigtail tube
  Arms: Puncture and Drainage

SUMMARY:
The acute peripancreatic fluid collections (AFPCs) is the most common complication in severe acute pancreatitis (SAP). There are controversies on optimal timing for drainage of APFCs in SAP. The early-stage percutaneous catheter drainage (PCD) of sterile peripancreatic fluid collections is questioned as a result of the major cause of secondary infection. The aim of the present randomized controlled trial is to compare the outcomes in terms of mortality, secondary infection of peripancreatic collections, organ failure, length of hospital/ICU stay and inflammatory biomarkers between the early-stage PCD of sterile AFPCs and conservative therapy.

DETAILED DESCRIPTION:
The AFPCs is the most common complication in SAP and debate continues regarding the appropriate timing for drainage of sterile APFCs in SAP patients. Some researchers have reported that the massive amounts of inflammatory mediators in the peripancreatic fluid may aggravate the inflammatory reaction and contribute to organ failure (OF) when liberated into the bloodstream by peritoneal absorption. Additionally, bacterial colonization of APFCs may lead to peritoneal abscess formation and sepsis. In a recent study, Wang et al. revealed that early-stage PCD effectively attenuated the peritoneal pressure and decreased the incidence of infection and OF. Finally, APFCs and secondary infection are considered major causes of alimentary tract hemorrhage. Based on these factors, prompt drainage of APFCs seems reasonable for patients in early SAP. In addition, unlike the original 1992 Atlanta classification guidelines (1992-AC), the revision of the 1992-AC by international consensus in 2012 (2012-RAC) highlighted the significance of persistent OF in the classification of SAP. To be exact, those patients diagnosed with SAP according to the 1992-AC without OF or with transient OF were reclassified as having mild AP (MAP) or moderate severity AP (MSAP) by the 2012-RAC. Therefore, many studies have reported changes in the treatment of SAP in the early stages since the 2012-RAC were published. We have retrospectively analyzed 361 patients with AP and found that the early-stage PCD of sterile APFCs in SAP-2012RAC patients can significantly reduce the mortality rate. However, on the contrary, the mainstream viewpoint holds that drainage is not necessary in the absence of infection of the peripancreatic fluid as the fluid can be absorbed completely and sterile PCD may increase the risk of iatrogenic infection. However, these mainstream views aimed at 1992-AC's SAP patients, which actually contain 2012-RAC's SAP and MSAP. Therefore, we hypothesized that the introduction of new AP severity classification methods may alter the indications for early aseptic drainage of AFPCs.

Does early PCD of sterile APFCs benefits patients or increases the secondary infection rate? In view of these problems, we plan to design a randomized controlled trial to compare the outcomes in terms of mortality, secondary infection of peripancreatic collections, organ failure, length of hospital/ICU stay and inflammatory biomarkers between the early-stage PCD of sterile AFPCs and conservative therapy. The aim of this prospective study is to investigate whether early PCD of sterile AFPCs can be used to SAP patients with AFPCs at early stage.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 years to 70 years; and
2. Pain characteristic of pancreatitis; and
3. Elevated serum lipase or amylase (≥3-fold upper normal range); and
4. Persistent organ failure >48 hours; and
5. Organ dysfunction occurred within 7 days after onset of pain; and
6. Presentation with a width of ≥2cm of APFCs in the peripheral tissues of the pancreas, the cyst of lesser omentum , or the paracolic sulci on CT image.

Exclusion Criteria:

1. History diseases of chronic organ dysfunction; or
2. Traumatic pancreatitis; or
3. Post-endoscopic retrograde cholangiopancreatography(ERCP) pancreatitis; or
4. Severe coagulopathy (INR>2); or
5. Severe thrombocytopenia (PLT≤50×109/L); or
6. No suitable route for puncturing; or
7. Pregnancy; or
8. Absent of informed consent from patient or representative.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-10-06 (Estimated); Primary Completion 2020-10-06 (Estimated); Study Completion 2020-10-06 (Estimated)

PRIMARY OUTCOMES:
Mortality | From date of admisstion until the date of in-hospital death or death within two weeks after discharging, whichever came first, assessed up to 1 year.
  Determine and compare the death rates in patients who are administered drainage and conservative therapy: Assess the total number of cases of death in each group (Treatment and control)

SECONDARY OUTCOMES:
Secondary infection of peripancreatic collections | From date of admisstion until the secondary infection of peripancreatic collections occurred, assessed up to 100 days
  Compare the secondary infection rates of peripancreatic collections in patients who are administered drainage and conservative therapy: Assess the total numbers of cases of secondary infection of peripancreatic collections in each group (Treatment and control)
New set of organ failure | From date of admisstion until new set of organ failure occurred, assessed up to 100 days
  Compare the new set of organ failure rates in patients who are administered drainage and conservative therapy: Assess the total numbers of cases of new set of organ failure in each group (Treatment and control)
Length of hospital/ICU stay | From date of admisstion until the patient is transfered to normal ward or discharge, whichever came first, assessed up to 1 year.
  Compare the length of hospital/ICU stay in patients who are administered drainage and conservative therapy
Aggressive procedures: open necrosectomy and minimally invasive retroperitoneal necrosectomy | From date of admisstion until the patient receives aggressive procedures, assessed up to 100 days
  Compare the aggressive procedures rates in patients who are administered drainage and conservative therapy.
Abdominal hemorrhage | From date of admisstion until the abdominal hemorrhage occurred, assessed up to 100 days
  Compare the abdominal hemorrhage rates in patients who are administered drainage and conservative therapy.
Digestive tract fistula | From date of admisstion until the Digestive tract fistula occurred, assessed up to 100 days
  Compare the digestive tract fistula rates in patients who are administered drainage and conservative therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- The second affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China